CLINICAL TRIAL: NCT00660608
Title: Conservation of Red Cell Mass, Oxygen Supply and Demand in Cardiac Surgery
Brief Title: Conservation of Red Cell Mass , Oxygen Supply and Demand in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Daxor Corporation (Industry)
Responsible Party: Mark Nelson, MD, VCU Medical Center
Other Study IDs: BVA 100
Record Dates: First submitted 2008-04-10; First posted 2008-04-17 (Estimated); Last update posted 2010-07-05 (Estimated); Status verified 2010-07

CONDITIONS: Coronary Artery Disease
Keywords: Transfusion regulation
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Fifty patients will be enrolled into the study. The purpose of the study is to investigate the relevance of Hct levels in determining need for transfusion during operations employing bypass as well as to test the hypothesis that, while HCt levels may decrease during surgery , red blood cell mass and tissue oxygenation remain fairly constant.

DETAILED DESCRIPTION:
Fifty adults( male or female-nonpregnant) whose weight is between 55-85 kg and are scheduled to undergo elective cardiac surgery with cardiopulmonary bypass for CABG or primary valve repair or replacement will be eligible. Patients with any history of abnormal bleeding disorders, urgent or emergent need for surgery, and combination surgeries will be excluded. Blood volume analysis will be performed with the DAXOR Blood Volume Analyzer BVA-100 System and the Volumex HSA I-131 radiopharmaceutical for use for determining circulating volume. Multiple timed sample points will be obtained. The DAXOR blood volume analyzer will batch samples and with input of patients height, weight, gender, time of draw, and corresponding Hct, calculate circulating total blood volume. We hypothesize that Total red cell mass is relatively well conserved( <20% decrease) during and immediately after surgery as long as major bleeding does not occur. We hypothesize that decrease in Hct during surgery are related to changes in circulating plasma volume. Total red cell O2 carrying capacity and O2 economics will be measured and it is also hypothesized that lowered Hct values, even as low as 15%, do not independently signal a tissue or whole body O2 deficit.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled to undergo elective Cabg or primary repair/replacement on bypass pump.
* Age 18 yrs or older
* Male or non pregnant female
* Weight between 55-85 kg.

Exclusion Criteria:

* Any known bleeding risks;
* Urgent or emergent surgery;
* Combined aortic and major vascular surgery;
* Pregnant women
* If participating in another study within last 90 days.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pre-OP, surgery clinics, inpatients
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Nelson, MD, Principal Investigator — VCU Medical Center; Carlos Arancibia, MD, Study Chair — VCU Medical Center
Locations (1):
- VCU Medical Center, Richmond, Virginia, United States